CLINICAL TRIAL: NCT01604954
Title: Does Food Labeling Influence Long-term Food Intake and Eating-related Variables in Women?
Acronym: MENU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laval University (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Véronique Provencher, Professeur sous octroi, Laval University
Allocation: Randomized | Model: Factorial | Masking: Single
Other Study IDs: INAF 2011-088
Record Dates: First submitted 2012-05-16; First posted 2012-05-24 (Estimated); Last update posted 2015-09-01 (Estimated); Status verified 2015-08

CONDITIONS: Obesity
Keywords: Food labeling
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Non-obese (Other): Non-obese women (BMI between 18.5 and 25 kg/m2)
  Interventions: Behavioral: Nutrient-label; Behavioral: Calorie-label; Behavioral: No label
- Obese (Other): Obese women (BMI between 30 and 40 kg/m2)
  Interventions: Behavioral: Nutrient-label; Behavioral: Calorie-label; Behavioral: No label

INTERVENTIONS:
Behavioral: Nutrient-label — A label indicating that the lunch they will eat is low in saturated fat and free from trans fat will be posted on the containers.
Behavioral: Calorie-label — A label indicating the amount of calories for a fixed serving plus information about daily caloric requirement ("The recommended daily caloric intake for an average adult is 2000 calories") will be posted on the containers.
Behavioral: No label — Lunches will be free from labels, so that no nutritional information will be provided to the participants(control group).

SUMMARY:
Weight management is a critical issue in developed countries where the prevalence of obesity is always increasing. While the mismatch of energy intake and energy expenditure is recognized as a leading cause of obesity, knowledge related to the determinants of healthy eating patterns are still an important issue to further address. Various nutrition-education campaigns have been implemented as a way to increase knowledge about healthy foods and facilitate the adoption of better eating behaviors. There is currently social and politic pressure on health authorities to increase availability of nutrition information as a way to tackle the obesity epidemic. Does nutrition information on food labels really contribute to improving dietary intake among the population and to helping them to better manage their body weight? Some evidence suggests that describing foods as healthy might have unintended enhancement effects on the acute amount of food and calories consumed. A better understanding of how and why nutrient and calorie labels influence acute and chronic intake is thus needed. This study investigate how providing nutritional information on food labels influences intake and eating-related variables over a 10-day period among women characterized by varying levels of adiposity. As it has never been investigated before, the present research will provide important knowledge on the long-term impacts of different food labeling strategies on the regulation of food intake. It will also help to determine whether weight status could influence the effects of perceptions about foods on intake, so that the investigators can identify individuals who mostly tend to overeat in specific situations. Consumer advocacy organizations are urging government to adopt policies regarding food labeling. Such research is thus of great relevance for the promotion of healthy body weight at the population level, as it will clearly contribute to assess how food labels should be used by health governing bodies in the context of the obesity epidemic.

DETAILED DESCRIPTION:
Much effort has been invested to educate Canadians about the importance of healthy eating and active living. Various food labeling strategies are currently used (e.g. nutrient-content claims approved by Health Canada), or strongly suggested (e.g. calorie information on restaurant menus), as tools to increase knowledge about healthy food choices and to help consumers make more so-called healthier choices. Does nutrition information on food labels really contribute to improve dietary intakes among the population? Some evidence does suggest that food labeling could influence consumer's choices and purchases. But, consumers remain confused about what healthy eating should be, and about how many calories they should be eating per day. Data suggest that only 50% of them truly understand and use food labels. Results regarding the impact of food labeling on intake are less convincing. We have recently shown that perceiving a snack food as healthy increased intake of that food by 35% in female students. Health halos promoted by nutrition information may lead consumers to draw misleading inferences from food labels. Considering current public pressure on health authorities to increased availability of nutrition information as a way to attack the obesity epidemic, long-term impact of food labeling strategies on food intake regulation represents a critical key issue that have not been yet investigated.

The general objective of the present research proposal is to investigate how providing nutritional information on food labels influences intake and eating-related variables over a 10-day period among women. We will more specifically:

1. Compare the impact of 1) nutrient quality and 2) calorie content food labels vs. "no label" condition on mean ad libitum intake and appetite sensations before/after meals over a 10-day period in women.
2. Examine how body weight (normal versus obesity) influences the impact of the nutrient quality and calorie content food labels on mean ad libitum intake and appetite sensations over a 10-day period in women.
3. Verify whether types of food labels influence attitudes towards meals offered (i.e. perceived healthiness, appropriateness, palatability) over a 10-day period in women.

ELIGIBILITY:
Inclusion Criteria:

* stable weight (± 2.5 kg) for at least 3 months prior to the study.
* BMI between 18.5 and 25 kg/m2 for the non-obese group and BMI between 30 and 40 kg/m2 for the obese group.

Exclusion Criteria:

* pregnant or lactating.
* aversion to the foods in the study.
* taking medication (e.g., corticosteroids,tricyclic antidepressants, atypical antipsychotics) and present chronic health problems (e.g.,food allergies, eating disorders, diabetes, hyperthyroidism) that could affect appetite measurements and food intake.

Ages: 25 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2011-08; Primary Completion 2013-05 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Mean ad libitum intake | Up to 2 years after the beginning of the study
  The mean amount per day of food eaten during the 10-day period (grams and calories).

SECONDARY OUTCOMES:
Appetite sensations | Up to 2 years after the beginning of the study
  Visual-analogue ratings of hunger and fullness(measured in millimeters) before and after each meal.

CONTACTS AND LOCATIONS:
Overall Officials: Véronique Provencher, Ph.D., Principal Investigator — Laval University
Locations (1):
- Institute of Nutraceuticals and Functionnal Foods (INAF), Québec, Quebec, Canada